CLINICAL TRIAL: NCT04015960
Title: Evaluation of the effectiVeness of an ADaptation of the Making It-Work Intervention in a French Environment-pilot
Brief Title: Inflammatory Arthritis and Difficulty at Work
Acronym: RENOIR
Status: Withdrawn | Type: Observational
Why Stopped: lack of ressources
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Anne-Christine Rat, Principal investigator, University of Lorraine
Other Study IDs: EVADE-pilot
Record Dates: First submitted 2019-06-27; First posted 2019-07-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — qualitative research and patient reported outcome measure (PROm) development

SUMMARY:
Despite biologic drugs and improvements of inflammatory arthritis (IA) treatment, many patients with inflammatory arthritis still face increased absenteeism, reduced at-work productivity and report difficulties working and having to give up their jobs. Such professional limitation generates psychological stress and it felt generally as a premature social ageing.

"Making-it-Work" is an intervention developed in English speaking Canada, which aims at enabling both patients and employers to intervene early during the course of inflammatory arthritis to reduce possible problems at work, and to prevent sick leave and future work disability in the long term and improve well-being at work.

As part of the EVADE (Evaluation of the effectiVeness of an ADaptation of the Making it-Work intervention in a French Environment) project which aims at evaluating the effectiveness of an adaptation of the "Making-it-Work" intervention, to the French environment, the investigators propose :

1. to identify the problems faced at work due to IA, patients needs, motivations to continue working and strategies helpful for maintaining employment.
2. to develop a questionnaire to assess difficulties at work, needs for adaptations and support and motivations to work of patients with inflammatory arthritis.

DETAILED DESCRIPTION:
The development of the patient-reported outcome (PRO) measure will comprise:

Step 1: Identifying themes and generating items by

* Conducting focus groups and/or individual semi-structured interviews with patients with IA to identify the problems faced at work due to the disease and identify strategies helpful for maintaining employment. Work characteristics, work environment, and social, economic factors and role of family members will receive specific attention.
* Conducting focus groups including patients with IA who stay at work despite the disease to identify their motivations and needs to stay at work.
* Conducting individual semi-structured interviews with health care professionals and professionals of the prevention and security at work
* Conducting the thematic analysis, following a general inductive approach

Step 2: Selecting items using a Delphi method using a panel of patients and health care professionals

Step 3: Items reconciliation and selection by an expert panel

Step 4: Cognitive debriefing of selected items (pre-test).

Step 5: Evaluate psychometric properties will follow the standards for assessing validity of a complex measurement scale, checking for truth, discrimination and feasibility ((Outcome Measures in Rheumatology (OMERACT) filter 2.0) according to the COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) check-list. Scale measurement properties will be assessed using Rasch measurement methods.

ELIGIBILITY:
1. Patients

   Inclusion Criteria:
   * Physician diagnosis of IA (rheumatoid arthritis, spondyloarthritis or psoriatic arthritis)
   * Age 18 to 65 years
   * Currently employed
   * Having concerns about their IA at work ("Do you have any concern about your arthritis affecting your ability to work now, or in the next five years?),

   Exclusion Criteria:

   • Sick leave of more than 3 years
2. Health care professionals (clinicians, nurses experts in therapeutic education, occupational physicians), a vocational counsellor, and professionals of the prevention and security at work, professionals from the pension insurance fund and health at work or professionals involved in accommodation of working conditions for disabled workers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory arthritis (rheumatoid arthritis, spondyloarthritis or psoriatic arthritis) with difficulties at work
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Problems faced at work due to IA, patients needs, motivations to continue working and strategies helpful for maintaining employment. | baseline
  focus groups and/or individual semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Christine Rat, MD, PhD, Principal Investigator — University of Lorraine; Isabelle Thaon, MD, PhD, Principal Investigator — University of Lorraine
Locations (1):
- Université Lorraine, Nancy, France

IPD SHARING:
Plan to Share IPD: No